CLINICAL TRIAL: NCT05395286
Title: Controlled Evaluation of Innovation Labs for Enhancing Collaboration Among Early Career Scholars in the CTSA Network
Brief Title: Innovation Labs to Enhance Collaboration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Larry Hawk, Ph.D., Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001360
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Collaboration Attitudes and Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Innovation Lab Group (Experimental): Randomized to attend the Innovation Lab
  Interventions: Behavioral: Innovation Lab
- Control Group (No Intervention): Randomized to NOT attend the Innovation Lab

INTERVENTIONS:
Behavioral: Innovation Lab — An Innovation Lab is a facilitated 5-day residential event designed to create novel, transdisciplinary and potentially transformative research ideas and proposals to address a specific grand challenge. Participants, along with a director, organizers, subject matter guides, and KI facilitators communally explore the problem space, generate a broad range of ideas, and form transdisciplinary teams to pursue research projects.
  Arms: Innovation Lab Group

SUMMARY:
We will conduct and evaluate the impact of two week-long Innovation Labs on collaboration attitudes and behavior among early career scholars. Applicants to each Innovation Lab will be screened and then randomized to either the Innovation Lab group or a control group.

DETAILED DESCRIPTION:
Building on the science of team science and preliminary work at the Buffalo and Vanderbilt CTSAs, we propose to work with our industry partner Knowinnovation to implement, assess, and disseminate an innovative and promising method for stimulating and nurturing new transdisciplinary research teams across the CTSA Program consortium: Innovation Labs. We will focus on early career investigators, have well-developed expertise, and will benefit from developing transdisciplinary collaborations. This work will further advance the field by taking a strong translational science approach to identify and test "best practices". To accomplish this, we will critically evaluate the impact of Innovation Labs in two preliminary randomized controlled trials (RCTs). In collaboration with NCATs and broad input from the CTSA network, we will develop a clinical and translational research grand challenge focus for each Innovation Lab. A diverse applicant pool of early career investigators invited from every CTSA hub in the consortium will be reviewed, and top applicants will be randomized to a 5-day residential Innovation Lab or "treatment as usual" control group (n=25/group/RCT). Measures of process and outcome will be collected from the application phase through 12-month follow-up and aggregated across the two RCTs. Given the preliminary nature of the work and an emerging consensus regarding the science of team science, primary outcomes will be measures of the depth and breadth of participants collaborative networks and attitudes towards collaboration, which we predict will be enhanced in the Innovation Lab group compared to the treatment as usual control group. We will also gather initial data on the degree to which Innovation Labs result in increased transdisciplinary collaborative output, including grant proposals, publications, and presentations. The significance of this work is clear: We aim to advance clinical and translational science by critically evaluating a potential "best practice" method for catalyzing collaborations and enhancing innovative translational research, a core goal of the CTSA Program. Our initial RCTs target an important segment of the workforce and begin the process of dissemination across the CTSA network, setting the stage for much broader implementation and impact.

ELIGIBILITY:
Inclusion Criteria:

Completion of application and baseline assessment.

For randomization:

* Faculty at a NIH CTSA hub institution or regional partner.
* Early stage investigators (NIH-defined as "within 10 years of completing his/her terminal research degree or is within 10 years of completing medical residency (or the equivalent)") who are emerging as independent scholars.
* Applications were reviewed for the above criteria and ranked by committee according to goodness of fit with the topic of the Innovation Lab, the quality and quantity of academic productivity and collaboration, and contribution to diversity of perspectives among Lab participants (e.g., biomedical and social/psychological, basic and applied). Top-ranked applicants were retained for randomization to the Innovation Lab group or control group.

All applicants (including 94 randomized ppts and 13 ppts who were not randomized) were encouraged to remain in the study and complete the follow-up assessments.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Change from Baseline MATRICx Benefits Scale | through study completion, an average of 15 months
  Self-report: Motivation Assessment for Team Readiness, Integration, and Collaboration (MATRICx; Mallinson, Lotrecchiano, et al., 2016) - Motivator scale
Change from Baseline MATRICx Threats Scale | through study completion, an average of 15 months
  Self-report: Motivation Assessment for Team Readiness, Integration, and Collaboration (MATRICx; Mallinson, Lotrecchiano, et al., 2016) - Threats scale
Change from Baseline Transdisciplinary Orientation Scale | through study completion, an average of 15 months
  Self-report: 12-item Transdisciplinary Orientation scale (TDO; Misra, Stokols, & Cheng, 2015)
Change from Baseline Collaboration Network Size | through study completion, an average of 15 months
  Objective size of network of collaborators from published articles on PubMed

SECONDARY OUTCOMES:
Change from Baseline Grants Submitted | through study completion, an average of 15 months
  Self-Reported Number of New Grants Submitted
ILab met goal - new collab | 3 months
  The Lab met the goal of forming new transdisciplinary collaborations (ILab group only)
ILab met goal - novel proposals | 3 months
  The Lab met the goal of developing novel grant proposals on long-lasting lifestyle interventions (ILab group only)
ILab - recommend | 3 months
  I would recommend an Innovation Lab to a colleague (ILab group only)
ILab - positive impact | 3 months
  My experience in the Innovation Lab will have a positive impact on my work at my home institution (ILab group only)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Derived] Hawk LW Jr, Murphy TF, Hartmann KE, Burnett A, Maguin E. A randomized controlled trial of a team science intervention to enhance collaboration readiness and behavior among early career scholars in the Clinical and Translational Science Award network. J Clin Transl Sci. 2023 Dec 14;8(1):e6. doi: 10.1017/cts.2023.692. eCollection 2024. PMID 38384923